CLINICAL TRIAL: NCT07394972
Title: Iron Absorption From Stabilized Lactoferrin: An Experimental Study in Iron Deficient Women (LOBSTER)
Brief Title: Absorption of Iron From Stabilized Lactoferrin: A Study in Women With Iron Deficiency
Acronym: LOBSTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nicole Stoffel (Other)
Responsible Party: Sponsor-Investigator, Nicole Stoffel, Prof. Dr., ETH Zurich
Organization: ETH Zurich (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: LOBSTER
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Iron Deficiency (Without Anemia)
Keywords: Lactoferrin; Iron Deficiency; Iron Absorption; Iron Fortification; Stable Iron Isotopes; Dietary Supplements; Iron Bioavailability
MeSH Terms: conditions — Iron Deficiencies | interventions — Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Ferrous sulfate + inhibitory meal (Active Comparator): 4 mg of iron (58Fe) as ferrous sulfate + inhibitory meal
  Interventions: Other: FeSO4 + meal-matrix
- Ferrous sulfate + native LF + inhibitory meal (Active Comparator): 4 mg iron (58Fe) as ferrous sulfate + native LF + inhibitory meal
  Interventions: Other: FeSO4 + native LF + meal-matrix
- Ferrous sulfate + encapsulated LF (sodium caseinate) + inhibitory meal (Experimental): 4 mg iron (57Fe) as ferrous sulfate + sodium caseinate-LF + inhibitory meal
  Interventions: Other: FeSO4 + NaCas-LF + meal-matrix
- Encapsulated LF-Fe (Sodium caseinate) + inhibitory meal (Experimental): 4 mg of iron (54Fe) encapsulated with LF in sodium caseinate + inhibitory meal
  Interventions: Other: NaCas-LF-Fe + meal-matrix
- Ferrous sulfate + encapsulated LF (low methoxy pectin) + inhibitory meal (Experimental): 4 mg of iron (54Fe) as ferrous sulfate + low methoxy pectin-LF + inhibitory meal
  Interventions: Other: FeSO4 + LMP-LF + meal-matrix
- Encapsulated LF-Fe (low methoxy pectin) + inhibitory meal (Experimental): 4 mg of iron (57Fe) encapsulated with LF in low methoxy pectin + inhibitory meal
  Interventions: Other: LMP-LF-Fe + meal-matrix
- Encapsulated LF-Fe (sodium caseinate) + water (Experimental): 100 mg of iron encapsulated with LF in sodium caseinate + water
  Interventions: Other: NaCas-LF-Fe + water
- Encapsulated LF-Fe (low methoxy pectin) + water (Experimental): 100 mg of iron encapsulated with LF in low methoxy pectin + water
  Interventions: Other: LMP-LF-Fe + water
- Ferrous sulfate + water (Active Comparator): 100 mg of iron as ferrous sulfate + water
  Interventions: Other: FeSO4 + water

INTERVENTIONS:
Other: FeSO4 + meal-matrix — Maize porridge with labelled ferrous sulfate (58Fe)
  Arms: Ferrous sulfate + inhibitory meal
Other: FeSO4 + native LF + meal-matrix — Maize porridge with labelled ferrous sulfate (58Fe) and lactoferrin
  Arms: Ferrous sulfate + native LF + inhibitory meal
Other: FeSO4 + NaCas-LF + meal-matrix — Maize porridge with labelled ferrous sulfate (57Fe) and in sodium caseinate encapsulated lactoferrin
  Arms: Ferrous sulfate + encapsulated LF (sodium caseinate) + inhibitory meal
Other: NaCas-LF-Fe + meal-matrix — Maize porridge with sodium caseinate-lactoferrin-Fe (intrinsically labeled with iron isotope 54)
  Arms: Encapsulated LF-Fe (Sodium caseinate) + inhibitory meal
Other: FeSO4 + LMP-LF + meal-matrix — Maize porridge with labelled ferrous sulfate (54Fe) and low methoxy pectin lactoferrin
  Arms: Ferrous sulfate + encapsulated LF (low methoxy pectin) + inhibitory meal
Other: LMP-LF-Fe + meal-matrix — Maize porridge with low methoxy pectin-lactoferrin-Fe (intrinsically labelled with iron isotope 57)
  Arms: Encapsulated LF-Fe (low methoxy pectin) + inhibitory meal
Other: NaCas-LF-Fe + water — Water with sodium caseinate-lactoferrin-Fe (intrinsically labelled with iron isotope 54Fe)
  Arms: Encapsulated LF-Fe (sodium caseinate) + water
Other: LMP-LF-Fe + water — Water with low methoxy pectin-lactoferrin-Fe (intrinsically labelled with iron isotope 57Fe)
  Arms: Encapsulated LF-Fe (low methoxy pectin) + water
Other: FeSO4 + water — Water with ferrous sulfate (labelled with iron isotope 58Fe)
  Arms: Ferrous sulfate + water

SUMMARY:
Lactoferrin (LF) is a natural iron-binding protein found in milk. It exists either in an iron-free state (apo-LF) or bound to iron (holo-LF). Whether LF binds iron to facilitate its absorption and/or to sequester iron from potential enteropathogens remains uncertain. However, while LF is a promising tool for treating iron deficiency, it is sensitive to heat during food processing and to the acidic environment of the human stomach. This degradation often causes LF to lose its functional properties before it can promote iron absorption effectively.

This study aims to evaluate whether encapsulating apo-LF (either alone or in combination with iron) can protect LF from digestion and enhance iron absorption. Using a randomized, crossover design, different encapsulation methods will be compared to determine which results in the highest iron absorption in women with iron deficiency.

All test compounds will be labeled with stable iron isotopes. Participants will consume the labeled compounds with a test meal or water in a randomized order, allowing for within subject comparisons. Fractional iron absorption will be measured 17 days after administration via the incorporation of labeled iron into red blood cells.

ELIGIBILITY:
Inclusion Criteria:

* Serum ferritin < 45 µg/L (iron depleted)
* Body weight < 70 kg
* Body mass index 18,5 - 24,9 kg/m2 (normal weight)
* Hemoglobin (Hb) > 120 g/L (nonanemic)
* C-reactive protein (CRP) < 5 mg/L (no inflammation)

Exclusion Criteria:

* Pregnant or lactating
* Strictly vegan
* Cigarette smoking (> 1 cigarette / week)
* Gastrointestinal or metabolic disorders affecting iron absorption or metabolism
* Use of medication known to affect iron metabolism (oral contraceptives are allowed)
* Intake of vitamin and mineral supplements in the 2 weeks before study start and during the study
* Blood transfusion, blood donation, or significant blood loss during the previous 4 months
* once enrolled, inability to follow study procedures or major illness
* Participation in another study with investigational drug within the 30 days preceding and during the present study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-02-17 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Fractional iron absorption (%) | Day 22
  Fractional iron absorption calculated as the percentage of the administered labelled iron dose incorporated into red blood cells. The calculation is based on the measured shift in iron isotope ratios in blood samples collected 17 days after intake compared to baseline.
Fractional iron absorption (%) | Day 43
  Fractional iron absorption calculated as the percentage of the administered labelled iron dose incorporated into red blood cells. The calculation is based on the measured shift in iron isotope ratios in blood samples collected 17 days after intake compared to day 22.
Fractional iron absorption (%) | Day 64
  Fractional iron absorption calculated as the percentage of the administered labelled iron dose incorporated into red blood cells. The calculation is based on the measured shift in iron isotope ratios in blood samples collected 17 days after intake compared to day 43.

SECONDARY OUTCOMES:
Hemoglobin (g/dL) | Day 1
  Iron status marker
Hemoglobin (g/dL) | Day 22
  Iron status marker
Hemoglobin (g/dL) | Day 43
  Iron status marker
Hemoglobin (g/dL) | Day 64
  Iron status marker
Serum Ferritin (µg/L) | Day 1
  Iron status marker
Serum Ferritin (µg/L) | Day 22
  Iron status marker
Serum Ferritin (µg/L) | Day 43
  Iron status marker
soluble Transferrin Receptor (mg/L) | Day 1
  Iron status marker
soluble Transferrin Receptor (mg/L) | Day 22
  Iron status marker
soluble Transferrin Receptor (mg/L) | Day 43
  Iron status marker
C-reactive protein (mg/L) | Day 1
  Chronic inflammation marker
C-reactive protein (mg/L) | Day 22
  Chronic inflammation marker
C-reactive protein (mg/L) | Day 43
  Chronic inflammation marker
Alpha-1-acid Glycoprotein (g/L) | Day 1
  Acute inflammation marker
Alpha-1-acid Glycoprotein (g/L) | Day 22
  Acute inflammation marker
Alpha-1-acid Glycoprotein (g/L) | Day 43
  Acute inflammation marker

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Ursula Stoffel, Prof., Principal Investigator — ETH Zurich
Locations (1):
- ETH Zurich, Laboratory of Clinical Biopharmacy, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No